CLINICAL TRIAL: NCT02468596
Title: Axonal Excitability Measured by QTRAC Technique in Patients With Anti-MAG Neuropathy
Brief Title: Use of QTRAC Technique to Measure Axonal Excitability in Anti-MAG Neuropathy
Acronym: EXCIMAG
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of recruitment
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AGN_2014-20
Record Dates: First submitted 2015-03-03; First posted 2015-06-11 (Estimated); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Peripheral Neuropathy Associated With Anti-myelin Associated Glycoprotein Antibodies (Anti-MAG Neuropathy)
Keywords: Axonal excitability; Neuropathy; QTRAC; anti-MAG; Electrophysiology

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patients (Experimental): Patients suffering from anti-MAG neuropathy
  Interventions: Other: QTRAC assessment; Other: Clinical assessment of peripheral nerve function

INTERVENTIONS:
Other: QTRAC assessment — Computerized analysis of the muscular response of musculus abductor pollicis brevis, to series of electrical stimulations of the median nerve
Other: Clinical assessment of peripheral nerve function — Clinometric assessment using RT-MRC, Martin vigirometer, RT-mISS, T25W, 9 hole peg test, and ataxia scale

SUMMARY:
The QTRAC method is an electrophysiological technique that assesses peripheral nerve axonal excitability, using computerized analysis of the muscular response of musculus abductor pollicis brevis, to series of electrical stimulations of the median nerve.

Because of its high sensitivity to small changes in axonal excitability, QTRAC may help improve the follow-up of patients suffering from peripheral neuropathy caused by anti-myelin-associated-glycoprotein antibodies (anti-MAG neuropathy), as axonal excitability is early affected in this disease.

The main aim of the study is to compare QTRAC results in anti-MAG neuropathy patients, with QTRAC results in healthy persons (matched for sex and age).

A secondary aim is to determine whether or not the disease's clinical severity (measured by quantitative clinical scores) is correlated with the results of the QTRAC and could be predicted by a model based on the several parameters measured in the QTRAC exploration.

100 anti-MAG neuropathy patients will undergo a QTRAC exploration and a thorough neurological examination with clinical scoring. The results will be compared with data (matched by sex and age) from the reference database on healthy subjects, that is provided with the QTRAC software.

The investigators expect to prove that QTRAC results are modified in anti-MAG neuropathy patients, and that the clinical severity of the disease can be predicted by a combination of QTRAC-measured parameters.

ELIGIBILITY:
Inclusion Criteria:

* Anti-MAG neuropathy (peripheral neuropathy and IgM monoclonal gammopathy with anti-MAG activity superior to 1000 BTU)

Exclusion Criteria:

* current treatment with a medication that modifies peripheral nerve excitability (e.g. anticonvulsivants)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2022-02 (Actual)

PRIMARY OUTCOMES:
QTRAC-measured refractority of the median nerve | Inclusion
  the duration of the refractory period of the median nerve (expressed in milliseconds) is automatically measured by the QTRAC system, using a series of double electrical stimulations (the first being supra-maximal and the second, sub-maximal) and progressively increasing the time between the two stimuli.

CONTACTS AND LOCATIONS:
Locations (8):
- France (8):
  - Service de Neurologie Hôpital Pellegrin, Bordeaux
  - Service de Neurologie Hôpital Henry Mondor, Créteil
  - Département de Neurologie Hôpital Roger Salengro, Lille
  - service de neurologie, CHU Limoges, Limoges
  - Service ENMG et pathologies Neuro Musculaires, Hôpital Neurologique Pierre Wertheimer, Lyon
  - Laboratoire des explorations fonctionnelles, Hôtel Dieu, Nantes
  - Service de Neurologie, Fondation Ophtalmologique Adolphe de Rothschild, Paris
  - Service de Neurologie CHU St Etienne, Saint-Etienne